CLINICAL TRIAL: NCT02256592
Title: Reconstitution of the Gut Microbiome to Reduce HIV-Associated Inflammation
Brief Title: Fecal Microbiota Transplantation in HIV
Acronym: FMT-HIV
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: American College of Gastroenterology (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Ma Somsouk, MD, MAS, Associate Professor, University of California, San Francisco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-12675
Record Dates: First submitted 2014-10-01; First posted 2014-10-03 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: HIV
Keywords: inflammation; microbiome; immune activation; fecal microbiota transplantation; dysbiosis
MeSH Terms: conditions — Inflammation; Dysbiosis | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fecal microbiota transplant (FMT) (Experimental): Donor fecal suspension will be delivered during colonoscopy to HIV+ individuals.
  Interventions: Drug: Fecal Microbiota

INTERVENTIONS:
Drug: Fecal Microbiota — 300 mL of fecal suspension from a healthy donor will be delivered during colonoscopy
  Other Names: stool transplant

SUMMARY:
Even in individuals treated for HIV, chronic immune activation persists and is associated with increased cardiovascular disease, liver disease, and mortality. HIV-infected individuals have imbalances in the community of intestinal microbes which is thought to contribute to increased and persistent inflammation. The purpose of this study is to examine the safety and durability of fecal microbiota transplant (FMT), the transfer of the bacterial community in stool from a healthy donor, in HIV+ individuals on anti-retroviral therapy. The study will also measure the effects of FMT on immune activation and inflammatory biomarkers in anti-retroviral treated HIV+ individuals.

DETAILED DESCRIPTION:
Despite antiretroviral therapy (ART), chronic immune activation persists and is a major driver of HIV disease progression and mortality among HIV-infected individuals. Importantly, persistent inflammation is strongly associated with increased cardiovascular events, accelerated liver disease, impaired immunologic recovery (e.g. low CD4 count, low CD4 to CD8 ratio), and mortality. Therefore, addressing persistent inflammation remains a major goal to restoring health in HIV-infected individuals.

Novel therapeutic strategies to decrease immune activation in treated HIV infection are needed. Marked disruption of the gut microbial composition, or dysbiosis, is characteristic of HIV-infected individuals and persists despite long-term ART. Recent studies demonstrate that the relative degree of gut microbiome disruption positively correlates with inflammatory markers (IL-6, kynurenine to tryptophan ratio). Microbial dysbiosis and its inflammatory consequences may be an attractive target for interventions to decrease immune activation in HIV+ individuals.

Fecal microbiome transplantation (FMT) has proven durable and successful as a therapeutic strategy against gut dysbiosis, such as in the treatment of recurrent Clostridium difficile infection, by restructuring the composition of the gut microbiome to resemble that of the healthy donor. FMT has an established record of safety with limited adverse effects, even in the context of immunocompromised and HIV-infected subjects. Donor selection and screening will be conducted by OpenBiome.

The objective of this phase I clinical trial is to establish the safety and durability of FMT in HIV+ individuals. The microbiome of recipients will be analyzed up to 8 weeks post FMT for evidence of engraftment from the donor microbiome. We will further examine the effect of FMT on markers of immune activation and inflammation in ART treated HIV-infected individuals.

ELIGIBILITY:
Inclusion Criteria:

1. HIV infected men and women 18-75 years of age.
2. On continuous anti-retroviral therapy for at least one year.
3. Undetectable viral load for at least one year.
4. Written informed consent obtained from the subject and ability of the subject to comply with the requirements of the study.

Exclusion Criteria:

1. CD4 T cell count less than 200 cells/mL.
2. Recent antibiotic use in the last 3 months.
3. Pregnant, breastfeeding, or unwilling to practice birth control during participation in the study.
4. Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.
5. Active GI symptoms: inflammatory bowel disease, abdominal pain, hematochezia, or other symptoms requiring medical evaluation and intervention.
6. Recent hospitalization or acute medical condition within preceding three months.
7. Severe comorbidities: cirrhosis, coagulopathy, heart failure, renal failure, and respiratory failure.
8. Testing positive for any of the stool screening test: Clostridium difficile toxin by PCR, routine bacterial culture for enteric pathogens (E coli, Salmonella, Shigella, Yersinia, Campylobacter), culture for Vibrio, fecal Giardia antigen, fecal Cryptosporidium antigen, acid-fast stain for Cyclospora and Isospora, ova and parasites, stool for Rotavirus via EIA.
9. History of anaphylaxis.
10. Major immunosuppressive medications (e.g., calcineurin inhibitors, exogenous glucocorticoids, biological agents, etc.) or systemic antineoplastic agents.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-10; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Safety of FMT in HIV-infected individuals on suppressive ART. | 0-24 weeks post-FMT
  Determine the proportion of individuals with AE/SAE. Record AE/SAE during FMT and post-FMT and determine if related to study procedure and graded for severity. Study stoppage criteria includes any serious AE that is at least possibly related to study treatment or any serious infection (e.g., bacteremia) in a sterile body site with an organism potentially acquired from the FMT product.
Engraftment of donor microbiome in HIV-infected individuals on suppressive ART. | 8 weeks post-FMT
  The weighted Canberra distance, which calculates community similarity based on shared OTU membership irrespective of phylogenetic relatedness, and weighted UniFrac which considers phylogenetic similarity of microbial communities, will both be applied to compare the microbiome of FMT recipients over time to those of the donor infusion sample.

SECONDARY OUTCOMES:
Plasma will be analyzed for changes in levels of markers of inflammation (e.g. IL-6, sCD14, kynurenine to tryptophan ratio) and CD4 and CD8 T cell activation | 8 weeks post-FMT
  pre-FMT and 8 weeks post-FMT.

CONTACTS AND LOCATIONS:
Overall Officials: Ma Somsouk, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco-San Francisco General Hospital, San Francisco, California, United States

REFERENCES:
- [Background] Duprez DA, Neuhaus J, Kuller LH, Tracy R, Belloso W, De Wit S, Drummond F, Lane HC, Ledergerber B, Lundgren J, Nixon D, Paton NI, Prineas RJ, Neaton JD; INSIGHT SMART Study Group. Inflammation, coagulation and cardiovascular disease in HIV-infected individuals. PLoS One. 2012;7(9):e44454. doi: 10.1371/journal.pone.0044454. Epub 2012 Sep 10. PMID 22970224
- [Background] Vujkovic-Cvijin I, Dunham RM, Iwai S, Maher MC, Albright RG, Broadhurst MJ, Hernandez RD, Lederman MM, Huang Y, Somsouk M, Deeks SG, Hunt PW, Lynch SV, McCune JM. Dysbiosis of the gut microbiota is associated with HIV disease progression and tryptophan catabolism. Sci Transl Med. 2013 Jul 10;5(193):193ra91. doi: 10.1126/scitranslmed.3006438. PMID 23843452